CLINICAL TRIAL: NCT01177761
Title: Effects of Exercise on Fracture Risk, Bone Mineral Density and Falls in Postmenopausal Women. The Long-term Erlangen Fitness and Prevention Study.
Brief Title: The Erlangen Fitness and Prevention Study (EFOPS).
Acronym: EFOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Behinderten- und Versehrten-Sportverband Bayern e.V. (Other); Netzwerk Knochengesundheit e.V. (Unknown)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Professor Dr. Wolfgang Kemmler, University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OFZ-EFOPS
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis; Osteopenia; Early Postmenopause
Keywords: Osteoporosis; exercise; fractures; Bone Mineral Density; CHD-risk
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity; Fractures, Bone | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Active Comparator): endurance,balance, power, resistance type exercise
  Interventions: Procedure: physical exercise
- sedentary control (No Intervention): Subjects were instructed to do not relevantly change their lifestyle

INTERVENTIONS:
Procedure: physical exercise — Two sessions/week, 50 weeks/year over 12 years of high intensity exercise training
  Arms: exercise

SUMMARY:
The study determines the long-term effect of exercise on osteoporotic fracture risk. Since actually no controlled supervised exercise study exceeds the time frame of 4 years, knowledge concerning the long-term effect of exercise on fractures and fracture-risk factors is scarce. Within the Erlanger Fitness and Osteoporosis Study (EFOPS, an ongoing controlled exercise study with currently 16 years of supervised exercise with 45-50 osteopenic, early-postmenopausal women in exercise and sedentary control group each, the investigators therefore focus on overall-fractures, Bone Mineral Density and falls.

ELIGIBILITY:
Inclusion Criteria:

* participants of the EFOPS-study,
* 12 years of exercise training according to the EFOPS-protocol (exercise).

Exclusion Criteria:

* medication and diseases affecting bone metabolism,
* inflammable diseases,
* cardiovascular diseases,
* start of relevant physical exercise programs beside the EFOPS protocol.

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 1998-10; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
overall-fractures (low-trauma) | 16 year follow-up
  As assessed by questionnaire and structured interview
Bone Mineral Density at Lumbar Spine and Proximal Femur | 16 year follow-up
  As assessed by Dual-Energy X-ray Absorptiometry (DEXA)

SECONDARY OUTCOMES:
10-year coronary heart disease (CHD) risk | 16 year follow-up
  As assessed by Framingham Risk Factor Calculator according to Wilson.
Metabolic Syndrome Z-Score | 16 year follow-up
  Metabolic Syndrome Z-Score Index according to Johnson

CONTACTS AND LOCATIONS:
Overall Officials: Willi A Kalender, PHD, MD, Study Chair — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Kemmler W, von Stengel S, Bebenek M, Engelke K, Hentschke C, Kalender WA. Exercise and fractures in postmenopausal women: 12-year results of the Erlangen Fitness and Osteoporosis Prevention Study (EFOPS). Osteoporos Int. 2012 Apr;23(4):1267-76. doi: 10.1007/s00198-011-1663-5. Epub 2011 May 28. PMID 21625881
- [Background] Kemmler W, von Stengel S. Dose-response effect of exercise frequency on bone mineral density in post-menopausal, osteopenic women. Scand J Med Sci Sports. 2014 Jun;24(3):526-34. doi: 10.1111/sms.12024. Epub 2012 Nov 28. PMID 23190199
- [Result] Engelke K, Kemmler W, Lauber D, Beeskow C, Pintag R, Kalender WA. Exercise maintains bone density at spine and hip EFOPS: a 3-year longitudinal study in early postmenopausal women. Osteoporos Int. 2006 Jan;17(1):133-42. doi: 10.1007/s00198-005-1938-9. Epub 2005 Aug 12. PMID 16096715
- [Result] Kemmler W, Engelke K, von Stengel S, Weineck J, Lauber D, Kalender WA. Long-term four-year exercise has a positive effect on menopausal risk factors: the Erlangen Fitness Osteoporosis Prevention Study. J Strength Cond Res. 2007 Feb;21(1):232-9. doi: 10.1519/R-20826.1. PMID 17313298
- [Result] Stengel SV, Kemmler W, Pintag R, Beeskow C, Weineck J, Lauber D, Kalender WA, Engelke K. Power training is more effective than strength training for maintaining bone mineral density in postmenopausal women. J Appl Physiol (1985). 2005 Jul;99(1):181-8. doi: 10.1152/japplphysiol.01260.2004. Epub 2005 Mar 3. PMID 15746294
- [Result] Kemmler W, Lauber D, Weineck J, Hensen J, Kalender W, Engelke K. Benefits of 2 years of intense exercise on bone density, physical fitness, and blood lipids in early postmenopausal osteopenic women: results of the Erlangen Fitness Osteoporosis Prevention Study (EFOPS). Arch Intern Med. 2004 May 24;164(10):1084-91. doi: 10.1001/archinte.164.10.1084. PMID 15159265
- [Result] Kemmler W, Wildt L, Engelke K, Pintag R, Pavel M, Bracher B, Weineck J, Kalender W. Acute hormonal responses of a high impact physical exercise session in early postmenopausal women. Eur J Appl Physiol. 2003 Sep;90(1-2):199-209. doi: 10.1007/s00421-003-0874-7. Epub 2003 Jul 9. PMID 14504954
- [Derived] Kemmler W, von Stengel S, Bebenek M, Kalender WA. Long-term exercise and risk of metabolic and cardiac diseases: the erlangen fitness and prevention study. Evid Based Complement Alternat Med. 2013;2013:768431. doi: 10.1155/2013/768431. Epub 2013 Jul 30. PMID 23983804
- See also: homepage Institute of Medical Physics University of Erlangen-Nürnberg — http://www.imp.uni-erlangen.de/